CLINICAL TRIAL: NCT05494034
Title: Yield of Implantable Cardiac Monitoring Device in Patients With Acute Ischemic Stroke.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National and Kapodistrian University of Athens (Other)
Responsible Party: Principal Investigator, Georgios Tsivgoulis, Professor & Chairman of Second Department of Neurology, School of Medicine, National & Kapodistrian University of Athens, "Attikon" University Hospital, Athens, Greece, National and Kapodistrian University of Athens
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: ICM07082022
Record Dates: First submitted 2022-08-07; First posted 2022-08-09 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: Stroke, Acute; Stroke; Stroke, Ischemic; Atrial Fibrillation
MeSH Terms: conditions — Stroke; Ischemic Stroke; Atrial Fibrillation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- implantable cardiac monitoring device ("Reveal LINQTM") (Experimental): All included patients will have long-term heart rate monitors (Reveal LINQ; Medtronic)
  Interventions: Device: Reveal LINQTM

INTERVENTIONS:
Device: Reveal LINQTM — implantable cardiac monitoring device ("Reveal LINQTM")

SUMMARY:
In this prospective cohort study, the investigators aim to investigate the incidence of ICM-detected AF in unselected ischemic stroke patients and its association with anticoagulation initiation and stroke recurrence.

DETAILED DESCRIPTION:
The study will be conducted among 4 tertiary centers of the cardioneurology network in the Athens Metropolitan area ("Attikon" University Hospital, Hippokrateion Hospital, "Georgios Gennimatas" General Hospital of Athens, NIMITS General Hospital of Athens). The Second Department of Neurology of the National and Kapodistrian University of Athens in "Attikon" University Hospital would also act as the coordinating center, comprising of a research group with significant clinical experience and numerous publications on PCM and stroke.

Consecutive acute ischemic stroke or TIA patients aged 40 years or older will be enrolled. Diagnosis of acute ischemic stroke will be based on clinical and neuroimaging evaluation [brain computed tomography (CT) scan or magnetic resonance imaging (MRI) scan]. Classification of stroke will be defined using the Trial of Org 10172 in Acute Stroke Treatment (TOAST) criteria. Patients with incomplete evaluation will be excluded, as previously described. Patients with known or newly detected AF at hospitalization will also be excluded. Stroke patients of all other etiologies presenting a HAVOC score ≥4 will be included in the study. Informed consent for participation in the study will be obtained from the patients or guardians of patients.

Sample size

Similar to previous studies, approximately 200 eligible patients will be recruited during a 4-year period (50 patients/year). Based on a retrospective analysis of the local stroke registry and considering the eligibility criteria for this study, it is estimated that at least 1,000 stroke patients should be screened in order to enroll 200 participants.

Baseline Evaluation

All demographics and vascular risk factors will be prospectively recorded for all patients using standard definitions. Complete hematological and biochemical screening, as well as immunological and thrombophilia testing where indicated, will be performed. A comprehensive stroke etiopathogenic evaluation will be performed, including neuroimaging with brain computed tomography (CT) and / or magnetic resonance imaging (MRI), vascular imaging (cervical duplex ultrasound, transcranial Doppler, CT angiography and / or magnetic resonance [MR] angiography), ECG, transthoracic and/or transesophageal echocardiography and 24-to-48-hour Holter-ECG monitoring.

In particular, among the risk factors assessed, the age at inclusion, the number of atrial premature beats during the Holter-ECG monitoring, the location of index ischemic stroke (cortical versus deep), the brain natriuretic peptide (BNP) values, the presence of left atrial enlargement as diagnosed according to the guidelines of the American Society of Echocardiography, the HAVOC score (hypertension, age, valvular heart disease, peripheral vascular disease, obesity, congestive heart failure, coronary artery disease), the CHA₂DS₂-VASc score and the HAS-BLED score will be also recorded.

Stroke severity on admission will be assessed with the use of the National Institute of Health Stroke Scale (NIHSS) score by certified neurologists. Stroke classification according to the Trial of Org 10172 in Acute Stroke Treatment (TOAST) will be performed by certified neurologists, comprising of five stroke subtypes: (a) large-artery atherosclerosis; (b) cardioembolism; (c) small-vessel occlusion; (d) stroke of other determined etiology; and (e) stroke of undetermined etiology.[23] Interventions All included patients will receive secondary stroke prevention treatment and long-term management depending on the stroke subtype and according to current guidelines.

All included patients will have long-term heart rate monitors (Reveal LINQ; Medtronic) implanted subcutaneously under local anesthesia in the left chest region. During monitoring time, all patients with ICM will be evaluated clinically and electrocardiographically for up to 3 years following hospital discharge. Follow-up visits will be performed at the stroke outpatient clinic of our institution by outpatient visits and / or telephone, as dictated by their clinical status and at the discretion of the treating vascular neurologist, as previously described. All ICM recordings will be reviewed by a specialized cardiologist. All included patients will also be monitored with annual MRI scans for up to 3 years.

In the cases of AF detection, anticoagulant treatment may be initiated at the discretion of the treating physician, considering that the CHA₂DS₂-VASc score of the included patients will be at least 2 points, due to the history of stroke.

Statistical Analysis

Continuous variables will be presented as mean ± SD (normal distribution) and as median with interquartile range (IQR, skewed distribution). Categorical variables will be presented as number of patients and the corresponding percentages. Statistical comparisons between two groups (AF detected and no-AF detected) will be performed using χ2 test, or in case of small expected frequencies, Fisher's exact test. Continuous variables will be compared by the use of the unpaired t test or Mann-Whitney U test, as indicated. Cumulative probabilities of AF by risk factors will be displayed according to the Kaplan-Meier method. Event rates will be compared using the log-rank statistic. Univariable and multivariable Cox proportional hazards regression models will be used to determine predictors of AF. Baseline variables having differences with a significance level <0.10 will be considered as candidates for multivariable time-to-event AF models. Statistical significance will be achieved if the p value is ⩽0.05 in multivariable logistic regression analyses. The Statistical Package for Social Science (SPSS Inc, Armonk, NY, USA; version 23.0 for Windows) will be used for statistical analyses.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive acute ischemic stroke or TIA patients aged 40 years or older will be enrolled.
* Diagnosis of acute ischemic stroke will be based on clinical and neuroimaging evaluation [brain computed tomography (CT) scan or magnetic resonance imaging (MRI) scan].
* Stroke patients of all other etiologies (apart AF) presenting a HAVOC score ≥4 will be included in the study.
* Informed consent for participation in the study will be obtained from the patients or guardians of patients.

Exclusion Criteria:

* Patients with incomplete evaluation will be excluded, as previously described. [22] -Patients with known or newly detected AF at hospitalization will also be excluded.
* Not providing informed consent.

Ages: 40 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-05-05 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2030-01-01 (Estimated)

PRIMARY OUTCOMES:
Paroxysmal Atrial Fibrillation > 120 seconds | 3 years
  the incidence of paroxysmal AF lasting 120 seconds or more in included patients evaluated with ICM.

SECONDARY OUTCOMES:
Paroxysmal Atrial Fibrillation > 6 minutes | 3 years
  B) the incidence of paroxysmal AF lasting 6 minutes or more in included patients evaluated with ICM.
anticoagulant initiation | 3 years
  C) the incidence of anticoagulant initiation among included patients.
recurrent ischemic strokes | 3 years
  D) the incidence of recurrent ischemic strokes in included patients evaluated with ICM at follow-up according to paroxysmal AF duration.
subclinical infracts on follow-up MRI | 3 years
  E) the incidence of subclinical infracts on follow-up MRI scans according to paroxysmal AF duration.
major hemorrhagic events | 3 years
  F) the incidence of major hemorrhagic events in included patients evaluated with ICM at follow-up according to paroxysmal AF duration.
stroke subtypes | 3 years
  G) the possible correlation between stroke subtypes and AF detection.
biomarkers | 3 years
  H) the possible correlation of several baseline risk factors (including age, stroke location, BNP values, number of atrial premature beats, left atrial enlargement, HAVOC, CHA₂DS₂-VASc and HAS-BLED scores) with AF detection.
comparison versus historical cohort | 3 years
  I) the comparison of the rates of recurrent stroke among the patients included in the present cohort and undergoing ICM versus historical controls that were evaluated by the standard 24-hour Holter-ECG monitoring.

CONTACTS AND LOCATIONS:
Locations (1):
- Second Department of Neurology, "Attikon" University Hospital, School of Medicine, National and Kapodistrian University of Athens, Athens, Greece, Athens, Greece